CLINICAL TRIAL: NCT01609998
Title: Open-Label, Dose-Escalation, Phase I Study of the Prime-Boost Investigational 2012/13 Seasonal Influenza DNA Vaccine, VRC-FLUDNA063-00-VP, Followed by the 2012/2013 Seasonal TIV Compared to TIV Prime-Boost in Children/Adolescents Ages 6-17
Brief Title: Seasonal Influenza DNA Vaccine & Seasonal Influenza Trivalent Inactivated Vaccine (TIV) in Children & Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VRC 702; VRC 702 (Other Grant/Funding Number: HHSN272201000049I)
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Influenza
Keywords: Influenza A (H1); Influenza A (H3); Influenza B; DNA Vaccine; Trivalent Inactivated Vaccine (TIV); Healthy Adolescents; Healthy Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1A (12-17yrs):1 mg DNA vaccine+TIV (Experimental): 2012/13 seasonal influenza DNA Vaccine (VRC-FLUDNA063-00-VP) at Day 0 and licensed 2012/13 TIV at Week 18±2 wks
  Interventions: Biological: Seasonal Influenza DNA vaccine; Biological: TIV
- Group 1B (6-11yrs):1 mg DNA vaccine+TIV (Experimental): 2012/13 seasonal influenza DNA Vaccine (VRC-FLUDNA063-00-VP) at Day 0 and licensed 2012/13 TIV at Week 18±2 wks
  Interventions: Biological: Seasonal Influenza DNA vaccine; Biological: TIV
- Group 2A (12-17yrs):4 mg DNA vaccine+TIV (Experimental): 2012/13 seasonal influenza DNA Vaccine (VRC-FLUDNA063-00-VP) at Day 0 and licensed 2012/13 TIV at Week 18±2 wks
  Interventions: Biological: Seasonal Influenza DNA vaccine; Biological: TIV
- Group 2B (6-11yrs):4 mg DNA vaccine+TIV (Experimental): 2012/13 seasonal influenza DNA Vaccine (VRC-FLUDNA063-00-VP) at Day 0 and licensed 2012/13 TIV at Week 18±2 wks
  Interventions: Biological: Seasonal Influenza DNA vaccine; Biological: TIV
- Group 3A: (12-17yrs): TIV+TIV (Active Comparator): Licensed 2012/13 TIV at Day 0 and Week 18±2 wks
  Interventions: Biological: TIV
- Group 3B: (6-11yrs): TIV+TIV (Active Comparator): Licensed 2012/13 TIV at Day 0 and Week 18±2 wks
  Interventions: Biological: TIV

INTERVENTIONS:
Biological: Seasonal Influenza DNA vaccine — VRC-FLUDNA063-00-VP is composed of 3 closed-circular DNA plasmids that encode for the hemagglutinin (HA) from the following 3 strains: A/California/04/2009 (H1); A/Victoria/361/2011 (H3), and B/Wisconsin/2010. DNA vaccine vials will be supplied at 4 mg/mL in single use vials. The 1 mg dosage is administered as 0.25 mL volume and the 4 mg dosage as a 1 mL volume.
  Other Names: VRC-FLUDNA063-00-VP; HA DNA Vaccine; Seasonal influenza trivalent DNA vaccine
  Arms: Group 1A (12-17yrs):1 mg DNA vaccine+TIV; Group 1B (6-11yrs):1 mg DNA vaccine+TIV; Group 2A (12-17yrs):4 mg DNA vaccine+TIV; Group 2B (6-11yrs):4 mg DNA vaccine+TIV
Biological: TIV — 2012/13 Seasonal Influenza Trivalent Inactivated Vaccine (TIV)
  Other Names: 2012/13 Seasonal Influenza Trivalent Inactivated Vaccine

SUMMARY:
This is a Phase I, dose escalation study in healthy adolescents and children (6-17 years) to evaluate the safety, tolerability, and immunogenicity of a prime-boost regimen of the 2012/2013 seasonal influenza DNA vaccine (HA DNA) followed by licensed 2012/2013 TIV vaccine. The comparator groups will receive licensed 2012/2013 TIV as prime and boost. The hypothesis is that the 2012/2013 HA DNA prime-TIV boost regimen will be safe and result in a broader and more durable immune response than is observed in age-matched comparator TIV-TIV groups.

DETAILED DESCRIPTION:
Vaccines are an effective way to prevent influenza infection. Each year the World Health Organization (WHO) and the U.S FDA recommend the influenza strains to include in the seasonal influenza vaccines. The licensed seasonal influenza vaccines are directed against 3 influenza virus strains: an influenza A H1N1, an influenza A H3N2, and an influenza B. The currently approved vaccines depend upon labor-intensive methods that limit manufacturing speed and capacity. Influenza vaccines that can be more rapidly produced and that induce stronger, broader and more persistent immune responses are a recognized public health need.

In this protocol we will evaluate an investigational seasonal influenza (HA DNA) vaccine in healthy adolescents and children (6-17 years). Some participants will receive HA DNA vaccine "prime" followed by licensed trivalent influenza vaccine (TIV) "boost" 18 weeks later. Other participants will receive two TIV injections 18 weeks apart. The results will be compared. The HA DNA vaccine and TIV are both directed at the 3 influenza strains selected for the 2012/2013 vaccines. Prior studies in adults of avian and seasonal influenza DNA vaccines have been completed. The DNA vaccinations were assessed as safe and well tolerated in adults. The immune response to avian influenza is augmented by DNA vaccine priming compared to two vaccinations with the inactivated avian influenza (H5N1)vaccine when the prime-boost interval is 12-24 weeks, but not when the prime-boost interval is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents aged 6 to 17 years inclusive and at least 20 kg in weight.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* Willing to have blood drawn 5 times over 42 weeks, including blood stored for research purposes.
* In good general health as assessed by medical history, vital signs and targeted physical examination; stable medical conditions that, in the opinion of the investigator, will not compromise the subject's participation in the study are acceptable.
* Capability of the legal adult representative of the minor to understand and comply with planned study procedures.
* Capability of the legal adult representative of the minor to provide written informed consent; assent will be obtained from the child/adolescent per requirements of the site institutional review board (IRB).
* For female adolescent of child-bearing potential (as defined by onset of menses): agrees to avoid becoming pregnant and to use effective method of contraception or practice abstinence for at least 21 day prior to the first study vaccine administration, until at least 4 weeks after the second study vaccination.
* Within 70 days prior to enrollment, hemoglobin within institutional normal limits, creatinine less than the upper limit of normal (ULN) and ALT ≤1.5 X ULN for respective age group.

Exclusion Criteria:

* History of Guillain-Barré syndrome.
* Active neoplasm or history of cancer.
* On-going immunosuppressive therapy or known to be immunosuppressed at the time of enrollment.
* Immunoglobulin (or similar blood product) therapy within 3 months prior to enrollment.
* Known to have HIV, hepatitis B or hepatitis C infection.
* Acute or chronic illness that, in the opinion of the investigator, precludes participation in the study.
* Developmental delay, neurologic disorder, or seizure disorder requiring ongoing medical management (note: history of febrile seizure is not an exclusion).
* Acute febrile and/or respiratory illness within one week prior to enrollment.
* Idiopathic urticaria within the year prior to enrollment.
* Allergy treatment with antigen injections, unless on maintenance schedule and allergy shots could be staggered with the study vaccinations, within 14 days (2 weeks) prior to enrollment.
* Asthma that is severe, unstable or required emergent care, urgent care, hospitalization or intubation during the previous two years or that is expected to require the use of oral, intravenous or high dose inhaled corticosteroids.
* Vaccination of any type within 2 weeks prior to enrollment or receipt of the 2012/2013 seasonal TIV any time prior to enrollment.
* Participating in or planning to begin participation in another investigational study during the projected time during which the subject would be in this study.
* Factors related to the legal representative that in the judgment of the investigator may affect the objective decision-making of the legal representative.
* For a female adolescent of child-bearing potential: breast-feeding, known pregnancy or positive urine or serum pregnancy test on day of study enrollment.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of solicited and unsolicited adverse events | 7 days after injection for solicited events; from 1st injection to study completion for unsolicited events
  Incidence is reported for solicited events for 7 days after each injection, for unsolicited adverse event (AE) of any severity for 28 days after each injection, and for serious adverse events or new chronic medical conditions through 24 weeks after the 2nd injection.
Mean change from baseline in safety laboratory measures | Day 28
  At day 28 (+/- 7 days) blood will be drawn prior to receiving the second injection to measure hemoglobin, creatinine, and alanine transaminase (ALT).
Number of subjects with influenza or influenza-like illnesses | Day 0 through 24 weeks post TIV boost (Day 294)
  Participants who experience at least one influenza or influenza-like illness will be counted.

SECONDARY OUTCOMES:
Proportion of subjects with either a baseline hemagglutination inhibition (HAI) titer <1:10 and post-vaccination HAI titer ≥1:40 or baseline HAI titer ≥1:10 and a minimum 4-fold rise in HAI titer for each of the 3 strains in the 2012/13 TIV at Week 22. | Week 22 (4 weeks after TIV boost)
  Blood is collected from all subjects at baseline and at 4 weeks after TIV boost(Week 22 +/- 7 days) for testing in an HAI assay for each of the 3 strains of influenza in the 2012/2013 TIV.
Proportion of subjects with a four-fold or greater rise from baseline (Day 0) and Week 22 in 2012/13 TIV specific H1, H3 and B neutralizing antibodies | Week 22 (4 weeks after TIV boost)
  Blood is collected from all subjects at baseline (Day 0) and 4 weeks after TIV boost (Week 22 +/- 7 days) for testing in a neutralizing antibody assays for 2012/13 strain-specific H1, H3 and B antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Barney Graham, S Graham, M.D., Ph.D., Study Director — Chief, Clinical Trials Core Vaccine Research Center, NIAID, NIH; Julie Ledgerwood, D.O., Study Chair — Deputy Chief, Clinical Trials Core Vaccine Research Center, NIAID, NIH
Locations (5):
- United States (5):
  - Emory Children's Center, Atlanta, Georgia
  - Saint Louis University - Doisy Research Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Gamble Program for Clinical Studies, Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Ledgerwood JE, Wei CJ, Hu Z, Gordon IJ, Enama ME, Hendel CS, McTamney PM, Pearce MB, Yassine HM, Boyington JC, Bailer R, Tumpey TM, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 306 Study Team. DNA priming and influenza vaccine immunogenicity: two phase 1 open label randomised clinical trials. Lancet Infect Dis. 2011 Dec;11(12):916-24. doi: 10.1016/S1473-3099(11)70240-7. Epub 2011 Oct 3. PMID 21975270
- [Background] Ledgerwood JE, Graham BS. DNA vaccines: a safe and efficient platform technology for responding to emerging infectious diseases. Hum Vaccin. 2009 Sep;5(9):623-6. doi: 10.4161/hv.8627. No abstract available. PMID 19779298
- [Result] Houser KV, Yamshchikov GV, Bellamy AR, May J, Enama ME, Sarwar U, Larkin B, Bailer RT, Koup R, Paskel M, Subbarao K, Anderson E, Bernstein DI, Creech B, Keyserling H, Spearman P, Wright PF, Graham BS, Ledgerwood JE; VRC 702 study team. DNA vaccine priming for seasonal influenza vaccine in children and adolescents 6 to 17 years of age: A phase 1 randomized clinical trial. PLoS One. 2018 Nov 2;13(11):e0206837. doi: 10.1371/journal.pone.0206837. eCollection 2018. PMID 30388160